CLINICAL TRIAL: NCT03559504
Title: Comparing EEG Patterns in Different Age Groups During General Anesthesia With Sevoflurane
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHoWMU-CR2017-03-216
Record Dates: First submitted 2018-04-03; First posted 2018-06-18 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2018-09

CONDITIONS: Anesthesia
Keywords: electroencephalography; general anesthesia; sevoflurane

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Group 1: Infant period: 1 month-1 year old
  Interventions: Drug: Sevoflurane Inhal Soln
- Group 2: Toddler period:1-3 years old
  Interventions: Drug: Sevoflurane Inhal Soln
- Group 3: Preschool age period:3-6 years old
  Interventions: Drug: Sevoflurane Inhal Soln
- Group 4: School age period:7-18 years old
  Interventions: Drug: Sevoflurane Inhal Soln
- Group 5: Adults:18-65 years old
  Interventions: Drug: Sevoflurane Inhal Soln
- Group 6: Elderly:65-80 years old
  Interventions: Drug: Sevoflurane Inhal Soln

INTERVENTIONS:
Drug: Sevoflurane Inhal Soln — Anesthesia will be induced by sevoflurane inhalation only with a tight-fitting facemask and a 4-l airflow of 100% oxygen. Sevoflurane inhalation will be adjusted in all age groups to maintain 1.0 MAC concentration

SUMMARY:
This study is being conducted to evaluate and assess the electroencephalography wave patterns in different age patients undergoing surgery under general anesthesia. The aim of our study is to compare the raw EEG waves in different age patients and analyze any changes in these patterns among various age groups and which of these groups will have the EEG signal of high-frequency waves or low frequency waves. Previous studies have shown that light sedation is often accompanied by decreasing posterior alpha waves and increasing the intensity of frontal/central beta waves. It is therefore of neuroscientific interest to assess whether the electroencephalographic correlates of sevoflurane-induced unconsciousness have different or similar frequency range among the age groups.

DETAILED DESCRIPTION:
EEG is a powerful tool that refers to the recording of the brain's spontaneous electrical activity along the scalp and it can be used to measure voltage fluctuations which result from ionic current flows within neurons found in the brain.The electroencephalogram is increasingly used to measure anesthetic drug effect on the central nervous system.The use of electroencephalographic monitors has been proven to decrease drug consumption during anesthesia and to lead to a faster recovery from anesthesia. Recently, the use of the Bispectral Index® (BIS®) monitor (Aspect Medical Systems, Newton, MA) has been shown to decrease the incidence of intraoperative awareness. Depth of anesthesia is frequently assessed using electroencephalogram processing systems, such as BIS and M-Entropy® (Datex-Ohmeda, Helsinki, Finland). The use of these monitors has been claimed to allow more accurate drug administration which has the theoretical benefit of avoiding phases of too light or too profound anesthesia and the associated risks of hemodynamic instability. Inadequate general anesthesia caused by under dosage causes intraoperative awareness whereas prolonged anesthesia increases the risk of postoperative complications because of over dosage. The most important factor that contributes to the inadequate general anesthesia is the current limited ability to determine the level of awareness. In this study, the investigators want to analyze the raw EEG waves under general anesthesia using sevoflurane of MAC 1.0 for different age groups from 0 to 80 years old. The relation between concentration of 1.0 MAC sevoflurane and raw EEG states in different age groups is relatively unstudied. In this prospective randomized study the investigators want to know if there is any correlation of brain waves under general anesthesia in different age groups. Given that the brain rapidly develops and undergoes significant changes from childbirth into adulthood, anesthesia induced EEG oscillations in children might differ from those of adults, and could vary significantly with age. Characterizing the structure of the EEG in relation to age would help establish the foundations for age-appropriate monitoring of brain states during general anesthesia and sedation in children. The investigators aimed to examine the effects of age on the EEG during general anesthesia, with sevoflurane as the sole hypnotic agent.

After arrival in the operating room, an intravenous line will be inserted into a large forearm vein, and standard monitors will be applied. Each patient will be continuously monitored by a 3-lead electrocardiogram, noninvasive arterial pressure, pulse oximetry, and end-tidal carbon dioxide concentration.

The induction of anesthesia will be the same in all age groups and will consist of sufentanil 0.2-0.3mcg/kg or fentanyl 1-2 mcg/kg before intubation and 0.2 mg/kg cisatracurium to facilitate intubation. Sevoflurane inhalation will be adjusted in all age groups to maintain 1.0 MAC concentration. After tracheal intubation, patients will be ventilated with a tidal volume of 6-8 ml/kg and the respiratory rate will be adapted to obtain an end-tidal carbon dioxide concentration of 30-35 mmHg.

ELIGIBILITY:
Inclusion Criteria:

* Patients age between 0 to 80 years old
* American Society of Anesthesiologists (ASA) I or II scheduled for minor surgeries under general anesthesia lasting less than 2 hours each.

Exclusion Criteria:

* Potential subjects with any neurological or psychiatric disease
* Relative or absolute contraindication to sevoflurane including pregnancy by patient self-report
* Any recent prescription or illicit medication use will be excluded
* Patients with a history of any disabling central nervous or cerebrovascular disease
* Patients who had received central nervous system-active drugs
* Patients with poor quality data, most likely because of poor electrode contact.

Ages: 1 Month to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 120 patients undergoing minor elective surgeries will be allocated in 6 age groups: 0-1 year old (infant period), 1-3 years old (toddler period), 3-6 years old (preschool age period), 7-18 years old (school age period), 18-65 years old (adults) and 65-80 years old (elderly).
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-09-05 (Actual); Study Completion 2018-09-05 (Actual)

PRIMARY OUTCOMES:
Electroencephalography among various ages. | The experiment will be carried out for 10 mins after induction of anesthesia and before beginning of the surgery.
  Monitoring the raw EEG changes among various ages. The raw EEG waves of each patient will be analyzed and the results will be compared among the groups. The investigators want to see if there is any difference of the EEG wave among the 6 groups under 1.0 MAC sevoflurane.

SECONDARY OUTCOMES:
Morphology of electroencephalogram during 1.0 (MAC) Minimum Alveolar Concentration sevoflurane | While the raw EEG wave is being recorded for a period of 10 mins, the investigators will adjust the concentration of sevoflurane bringing it to 1.0 MAC.
  The investigators will analyze raw EEG waves from 0 year old to 80 years old. The subjects will be divided into 6 groups according to their respective age. Sevoflurane will be maintained at 1.0 MAC for each age groups.

CONTACTS AND LOCATIONS:
Locations (1):
- The second Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University and Yuying Children's Hospital of Wenzhou Medical University, Zhejiang, Zhejiang, China

DOCUMENTS (2):
  • Study Protocol (2018-06-27): https://cdn.clinicaltrials.gov/large-docs/04/NCT03559504/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-27): https://cdn.clinicaltrials.gov/large-docs/04/NCT03559504/SAP_001.pdf